CLINICAL TRIAL: NCT02731794
Title: Inflammatory Response and Clinical Outcome After On-pump Beating Coronary Artery Bypass Grafting Using Left Ventricular Assist Versus Biventricular Assist in Patients With Severe Left Ventricle Dysfunction
Brief Title: On-pump Beating Coronary Artery Bypass Grafting by Ventricular Assist
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Principal Investigator, Jian Zhao, associate professor, Henan Institute of Cardiovascular Epidemiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HenanICE201602
Record Dates: First submitted 2016-03-20; First posted 2016-04-08 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Bypass
Keywords: cardiopulmonary bypass; coronary artery bypass grafting; inflammatory response; cardiac dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LVA group (Experimental): LVA group: left ventricular assist group.
  Interventions: Device: left ventricular assist
- BiVA group (Active Comparator): BiVA group: Biventricular assist group.
  Interventions: Procedure: Biventricular assist

INTERVENTIONS:
Device: left ventricular assist — In left ventricular assist group, 100 IU/kg heparin was given to activated clotting time (ACT) greater than 180 seconds. A 22 French arterial cannula (Maquet, Irrlingen, Germany) was introduced into the ascending aorta, and a 26 French cannula (Eurosets, Medolla, Italy) into the left atrium and advanced into the left ventricle. The two cannulas are directly connected through a short, heparin-coated circuit to a centrifuge pump (Maquet, Getinge Group, Germany). A flow of 1.0 to 4.0 L/min/m2 is obtained and mean blood pressure was maintained 55-75 mm Hg. Note: Both LVA group and BiVA group have the operative protocols itself,includes different prime fluid and cannula pathway. The investigators think it is inapplicable to assign the different operative protocols to the Treatment Arm.
  Arms: LVA group
Procedure: Biventricular assist — In biventricular assist group, the patients were routinely heparinized with a dose of 300 IU/kg heparin to ACT greater than 480 seconds. Cardiopulmonary bypass with a centrifuge pump (Maquet, Getinge Group, Germany) was established by 22 French aortic cannulation and 34 French two-stage venous cannula through the right atrial appendage. The extracorporeal circuit was primed with 2000 mL of lactated Ringer's solution, albumin, 25% mannitol and 5% NaHCO3. The flow was 1.0 to 4.0 L/min/m2 and mean blood pressure was maintained 55-75 mm Hg.
  Arms: BiVA group

SUMMARY:
The investigators designed the randomized prospective study to evaluate the differences of inflammatory response and clinical outcome after on-pump beating coronary artery bypass grafting undergoing left ventricular assist versus biventricular assist in patients with severe left ventricle dysfunction.

DETAILED DESCRIPTION:
Off-pump coronary artery bypass grafting (CABG) tends to have a lower incidence of postoperative complications and remarkable advantages in terms of hospital stay. However, some drawbacks include higher rates of incomplete revascularization and the hemodynamic deterioration during manipulation of the heart, more occurring in the cases of posterolateral anatomical constraints and cardiac dysfunction. It leads to urgent conversion to extracorporeal circulation (ECC) and increases the mortality. Although conventional ECC with cardioplegia arrest provides bloodless immovable field, intense systemic inflammatory response may contribute to hemodynamic unstability especially in patients already with severe cardiac dysfunction.

On-pump beating CABG, as a more comprehensive approach, not only facilitates stable hemodynamics and complete revascularization, but also supports myocardial lymphatic flow balance and decreases interstitial myocardial edema in the beating state. Especially in the high-risk patients,some findings suggested that off-pump CABG should be converted to on-pump beating CABG without hesitation, avoiding hemodynamic collapse and even catastrophic outcomes. Some investigators intentionally planned on-pump beating CABG aiming to some patients with severe left ventricle dysfunction. Furthermore, on-pump beating CABG with ECC assistance in a high-risk subgroup is also an acceptable trade-off between conventional cardioplegia and off-pump operations.

The above-mentioned ECC results about on-pump, beating-heart CABG pay much attention to the biventricular assist (BiVA). Nonetheless, much evidence also reveals that BiVA triggers an intense inflammatory response due to extracorporeal membrane lung and circuit line. Comparatively speaking, single left ventricular assist (LVA), with shorter circuit line, less priming volume and free of extracorporeal membrane lung, theoretically should reduce the inflammatory response and relative complications. As a result, aiming to the high-risk patients with severe left ventricle dysfunction, who need ECC assistance (BiVA or LVA), the investigators designed the randomized prospective study to evaluate: 1) the differences in myocardial injury as expressed by cardiac Troponin I(cTnI) and in inflammatory response by C-reactive protein (CRP), 2) the differences in the early postoperative outcomes including graft number, incidence of atrial fibrillation, in-hospital mortality and ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe left ventricle dysfunction with an ejection fraction (EF)≤40%, being scheduled for revascularization.

Exclusion Criteria:

* myocardial infarction within the preceding 4 weeks
* severe valve disease requiring valve replacement
* cardiac reoperations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-05; Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Changes of C-reactive protein (CRP) | up tp 72 hours
  Serial blood samples for inflammatory response of CRP were collected at the following time points: 1: induction of anesthesia, 2: upon termination of cardiopulmonary bypass (CPB), 3: 6 hours postoperatively, 4: 24 hours postoperatively, 5: 48 hours postoperatively, 6: 72 hours postoperatively.

SECONDARY OUTCOMES:
Incidence of atrial fibrillation | 10 days
  from ICU admission to discharge
Durations of mechanical ventilation | 10 days
The number for transfused packed red cells | up to 10 days
  measured by milliliter from ICU admission to discharge
Partial oxygen pressure/inspired oxygen fraction (P/F) | up tp 10 days
Cardiac Troponin I (cTnI) | up to72 hours
  Serial blood samples for cTnI were collected at the following time points: 1: induction of anesthesia, 2: upon termination of CPB, 3: 6 hours postoperatively, 4: 24 hours postoperatively, 5: 48 hours postoperatively, 6: 72 hours postoperatively.
In-hospital mortality | up to 10 days
  from ICU admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoyun Cheng, MD, Study Director — Henan Provincial People' Hospital
Locations (1):
- Henan Provincial People' Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lim E, Drain A, Davies W, Edmonds L, Rosengard BR. A systematic review of randomized trials comparing revascularization rate and graft patency of off-pump and conventional coronary surgery. J Thorac Cardiovasc Surg. 2006 Dec;132(6):1409-13. doi: 10.1016/j.jtcvs.2006.08.012. PMID 17140968
- [Result] Urso S, Sadaba JR, Pettinari M. Impact of off-pump to on-pump conversion rate on post-operative results in patients undergoing off-pump coronary artery bypass. Interact Cardiovasc Thorac Surg. 2012 Feb;14(2):188-93. doi: 10.1093/icvts/ivr071. Epub 2011 Nov 28. PMID 22159253
- [Result] Fujii T, Watanabe Y, Shiono N, Kawasaki M, Yokomuro H, Ozawa T, Hamada S, Masuhara H, Teramoto T, Hara M, Katayanagi T, Sasaki Y, Koyama N. Assessment of on-pump beating coronary artery bypass surgery performed after introduction of off-pump approach. Ann Thorac Cardiovasc Surg. 2006 Oct;12(5):324-32. PMID 17095974
- [Result] Erkut B, Dag O, Kaygin MA, Senocak M, Limandal HK, Arslan U, Kiymaz A, Aydin A, Kahraman N, Calik ES. On-pump beating-heart versus conventional coronary artery bypass grafting for revascularization in patients with severe left ventricular dysfunction: early outcomes. Can J Surg. 2013 Dec;56(6):398-404. doi: 10.1503/cjs.018412. PMID 24284147
- [Result] Mazzei V, Nasso G, Salamone G, Castorino F, Tommasini A, Anselmi A. Prospective randomized comparison of coronary bypass grafting with minimal extracorporeal circulation system (MECC) versus off-pump coronary surgery. Circulation. 2007 Oct 16;116(16):1761-7. doi: 10.1161/CIRCULATIONAHA.107.697482. Epub 2007 Sep 17. PMID 17875971
- [Result] Al Jaaly E, Chaudhry UA, Harling L, Athanasiou T. Should we consider beating-heart on-pump coronary artery bypass grafting over conventional cardioplegic arrest to improve postoperative outcomes in selected patients? Interact Cardiovasc Thorac Surg. 2015 Apr;20(4):538-45. doi: 10.1093/icvts/ivu425. Epub 2014 Dec 21. PMID 25535178
- [Result] Stassano P, Di Tommaso L, Monaco M, Iesu S, Brando G, Buonpane S, Ambrosio G, Di Benedetto G, Pepino P. Myocardial revascularization by left ventricular assisted beating heart is associated with reduced systemic inflammatory response. Ann Thorac Surg. 2009 Jan;87(1):46-52. doi: 10.1016/j.athoracsur.2008.07.098. PMID 19101266
- [Result] Gulcan O, Turkoz R, Turkoz A, Caliskan E, Sezgin AT. On-pump/beating-heart myocardial protection for isolated or combined coronary artery bypass grafting in patients with severe left ventricle dysfunction: assessment of myocardial function and clinical outcome. Heart Surg Forum. 2005;8(3):E178-82; discussion E183. doi: 10.1532/HSF98.20041166. PMID 15937002
- [Result] Ferrari E, Stalder N, von Segesser LK. On-pump beating heart coronary surgery for high risk patients requiring emergency multiple coronary artery bypass grafting. J Cardiothorac Surg. 2008 Jul 2;3:38. doi: 10.1186/1749-8090-3-38. PMID 18597673
- [Result] Folliguet TA, Philippe F, Larrazet F, Dibie A, Czitrom D, Le Bret E, Bachet J, Laborde F. Beating heart revascularization with minimal extracorporeal circulation in patients with a poor ejection fraction. Heart Surg Forum. 2002;6(1):19-23. doi: 10.1532/hsf.992. PMID 12611727